CLINICAL TRIAL: NCT01470170
Title: The Optimal Regimen of Alfentanil in Propofol Sedative Fibro-bronchoscopy：a Prospective Randomized, Double-blind, Placebo-controlled Trial
Brief Title: Regimen of Alfentanil in Propofol Sedative Fibro-bronchoscopy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Chung-Hsing, Hsieh, Chief of Medical Intensive Care Unit, Department of Internal Medicine, Chang-Gung Memorial Hospital, Taipei, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 99-1538A3
Record Dates: First submitted 2011-10-27; First posted 2011-11-11 (Estimated); Results first posted 2015-08-13 (Estimated); Last update posted 2015-08-13 (Estimated); Status verified 2015-08

CONDITIONS: Hypoxemia
Keywords: Sedative bronchoscope; Alfentanil doses; Propofol; Targeted controlled infusion; Hypoxemia
MeSH Terms: conditions — Hypoxia | interventions — Alfentanil; Saline Solution; Propofol

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (5):
- Group1 (Experimental): Alfentanil 2.5μg/kg before propofol
  Interventions: Drug: Alfentanil; Drug: Normal saline; Device: Targeted controlled infusion; Drug: Propofol
- Group2 (Experimental): Alfentanil 5μg/kg before propofol
  Interventions: Drug: Alfentanil; Drug: Normal saline; Device: Targeted controlled infusion; Drug: Propofol
- Group 3 (Experimental): Alfentanil 2.5μg/kg two minutes before propofol
  Interventions: Drug: Alfentanil; Drug: Normal saline; Device: Targeted controlled infusion; Drug: Propofol
- Group 4 (Experimental): Alfentanil 5μg/kg two minutes before propofol
  Interventions: Drug: Alfentanil; Drug: Normal saline; Device: Targeted controlled infusion; Drug: Propofol
- Group 5 Control (Placebo Comparator): propofol alone
  Interventions: Drug: Normal saline; Device: Targeted controlled infusion; Drug: Propofol

INTERVENTIONS:
Drug: Alfentanil — Give Alfentanil before TCI Propofol sedative bronchoscope
  Arms: Group 3; Group 4; Group1; Group2
Drug: Normal saline — Normal Saline (placebo comparator) was given in equivalent amount of alfentanil dosage in each arm, for double blinded purpose.
Device: Targeted controlled infusion — The Propofol dosage was according to the effect site concentration to reach OAAS-3 ( loss of conscious), using Schneider model
Drug: Propofol — The Propofol dosage is according to the effect site concentration to reach OAAS-3 ( loss of conscious), using TCI Schneider model during the whole procedure of bronchoscope

SUMMARY:
Alfentanil (Alf) is used in combination with Propofol (Pro) in fiber-bronchoscopy and in many other conscious sedation procedures. Alf and Pro have the characteristic of rapid anesthetic onset and quick recovery, synergic sedative effect and unwanted side effects too. However, the amount of Alf needed in combination with Pro for induction and the timing of administration was no standardized. The investigators designed this study to evaluate the optimal regimen, dose and timing of Alf in Target-Controlled infusion (TCI) of Pro for flexible bronchoscopy sedation, and also to evaluate the influence of variable regimen of Alf and Pro on hypoxemia, hypotension, cough severity, and Pro injection related pain.

DETAILED DESCRIPTION:
Alfentanil (Alf) is used in combination with Propofol (Pro) in fiber-bronchoscopy and in many other conscious sedation procedures. Alf and Pro have the characteristic of rapid anesthetic onset and quick recovery, synergic sedative effect and unwanted side effects too. However, the amount of Alf needed in combination with Pro for induction and the timing of administration was no standardized. The investigators designed this study to evaluate the optimal regimen, dose and timing of Alf in Target-Controlled infusion (TCI) of Pro for flexible bronchoscopy sedation.

Method: patients will be enrolled and assigned randomly into five groups. In group 1, normal saline two minutes before and Alf 2.5μg/kg before Pro were given; In group 2, normal saline two minutes before and Alf 5μg/kg before Pro were given; In group 3, Alf 2.5μg/kg two minutes before and normal saline before Pro were given; In group 4: Alf 5μg/kg two minutes before and normal saline before Pro were given; in group 5, normal saline two minutes and before Pro were given.

Concentration of effect site to loss of consciousness (LOC), dose of Pro to LOC, and induction time of variable regimen, as well as hypoxemia, hypotension, cough severity, and Pro injection related pain will be recorded and analyzed.

ELIGIBILITY:
Inclusion Criteria:

* patients who required elective sedative bronchoscopy

Exclusion Criteria:

* any physical, psychiatric, social problem that avoid from conscious level evaluation,
* hypersensitivity or allergy to Propofol, Alfentanil
* severe chronic obstructive pulmonary disease (forced expiratory volume in 1 s ,50% of predicted value, or requirement for oxygen therapy)
* unstable haemodynamic status (defined as a heart rate < 60 or ≧ 120 bpm and/or
* a systolic blood pressure (SBP) < 100 or ≧ 180 mmHg)
* predictable difficult upper airways (Mallampati classification score of IV)
* severe obstructive sleep apnea with apnea hypopnea index (AHI) > 45
* Body mass index (BMI) more than 42 in male and 35 in female
* renal insufficiency
* liver cirrhosis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 173 (Actual)
Dates: Start 2010-10; Primary Completion 2011-09 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chung Hsing Hsieh, M.D., Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Taipei, Taiwan

RESULTS

PARTICIPANT FLOW:
Groups:
- Group1: Alfentanil 2.5μg/kg immediately before TCI propofol administration
- Group2: Alfentanil 5μg/kg immediately before TCI propofol administration
- Group 3: Alfentanil 2.5μg/kg two minutes before TCI propofol administration
- Group 4: Alfentanil 5μg/kg two minutes before TCI propofol administration
- Group 5 Control: TCI propofol administration alone
Period: Overall Study
Arm/Group | Group1 | Group2 | Group 3 | Group 4 | Group 5 Control
Started | 34 | 35 | 34 | 36 | 34
Completed | 34 | 35 | 34 | 36 | 34
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group1: alfentanil 2.5ug/kg immediately before propofol
- Group 2: alfentanil 2.5ug/kg two minutes before propofol
- Group 3: alfentanil 5ug/kg immediately before propofol
- Group 4: alfentanil 5ug/kg two minutes before propofol
- Group 5/ Control: Propofol alone
- Total: Total of all reporting groups
Arm/Group | Group1 | Group 2 | Group 3 | Group 4 | Group 5/ Control | Total
Number analyzed (Participants) | 34 | 35 | 34 | 36 | 34 | 173
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.3 (11.9) | 60.3 (15.8) | 58.8 (13.0) | 60.9 (13.9) | 62.2 (11.1) | 60.5 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 13 | 17 | 12 | 13 | 70
  Male | 19 | 22 | 17 | 24 | 21 | 103
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 23.7 (2.4) | 23.5 (3.4) | 23.8 (4.5) | 23.5 (3.3) | 23.2 (3.7) | 23.54 (3.5)
American Society of Anaethesiology Physical Status Score [Number; unit: participants]
  1 Normally healthy | 19 | 23 | 23 | 19 | 24 | 108
  2 Discrete systemic disease | 7 | 5 | 7 | 10 | 6 | 35
  3 Serious, non-incapacitating systemic disease | 8 | 7 | 4 | 7 | 4 | 30
Mallampati Score [Number; unit: participants]
  I: soft palate, uvula, fauces, pillars visible | 4 | 6 | 4 | 5 | 7 | 26
  II: soft palate, uvula, fauces visible | 16 | 13 | 14 | 10 | 12 | 65
  III: soft palate, base of uvula visible | 14 | 16 | 16 | 21 | 15 | 82
Regular use of opioid [Number; unit: participants] — use of opioid related medication for more than 5 days per week
  participants | 1 | 1 | 1 | 0 | 0 | 3
Regular use of sedation drugs [Number; unit: participants] — use of sleeping pill or sedative medication for more than 5 days per week
  participants | 3 | 2 | 4 | 5 | 3 | 17
Alcohol use [Number; unit: participants] — alcohol drinking for more than 5 days per week
  participants | 3 | 4 | 1 | 5 | 4 | 17
smoking status [Number; unit: participants]
  never | 20 | 18 | 21 | 19 | 20 | 98
  current | 7 | 12 | 8 | 11 | 6 | 44
  ex- | 7 | 5 | 5 | 6 | 8 | 31
heart rate [Mean (Standard Deviation); unit: beats/min] | 80.3 (15.5) | 78.1 (12.6) | 73.9 (14.2) | 80.3 (14.5) | 80.2 (11.4) | 78.6 (14.4)
SBP [Mean (Standard Deviation); unit: mmHg] | 147.1 (24.3) | 139.9 (20.5) | 139.2 (20.8) | 142.4 (21.5) | 145.8 (20.5) | 142.9 (21.5)
DBP [Mean (Standard Deviation); unit: mmHg] | 80.8 (12.7) | 78.7 (13.5) | 76.9 (11.8) | 79.5 (12.1) | 80.2 (11.4) | 79.2 (12.2)
SpO2 [Mean (Standard Deviation); unit: percentage of saturation] | 98.8 (1.5) | 98.6 (1.5) | 99.0 (1.4) | 99.2 (1.3) | 99.1 (1.5) | 98.9 (1.4)

OUTCOME MEASURES:

1. Primary Outcome: Effect Site Concentration When Conscious Level Reaches OAAS-3
Description: After the administration of alfentanil and propofol, the effect site concentration was recorded at the time when the consciousness level reaches observer assessment of alertness and sedation scale 3 (OAAS-3). The effect site concentration is the concentration of drug propofol in brain calculated by TCI using Schnider model.
Time Frame: All participants wil be follow for the duration of bronchoscope room stay, an expect average of 2 hours
Measure: Mean (Standard Deviation); unit: ug/ml
Groups:
- Group 5 /Control: Propofol alone
Arm/Group | Group1 | Group 2 | Group 3 | Group 4 | Group 5 /Control
Number analyzed (Participants) | 34 | 35 | 34 | 36 | 34
ug/ml | 2.3 (0.4) | 2.2 (0.4) | 2.5 (0.4) | 2.2 (0.5) | 2.6 (0.4)

2. Primary Outcome: Propofol Dose Needed to Reach Conscious Level OAAS-3
Description: After the administration of Alfentanil and Propofol, the Propofol dose needed to reach conscious level of observer assessment of alertness and sedation scale 3 (OAAS-3) will be recorded.
Time Frame: All participants wil be follow for the duration of bronchoscope room stay, an expect average of 2 hours
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Group1 | Group 2 | Group 3 | Group 4 | Group 5 /Control
Number analyzed (Participants) | 34 | 35 | 34 | 36 | 34
mg | 67.8 (56.2) | 56.4 (29.2) | 75.3 (37.1) | 54.8 (29.0) | 76.3 (31.9)

3. Primary Outcome: Induction Time, Time Period That Will be Required for Conscious Level to Reach OAAS-3
Description: After the administration of Alfentanil and Propofol, the time period required to reach conscious level OAAS-3 will be recorded.
Time Frame: All participants wil be follow for the duration of bronchoscope room stay, an expect average of 2 hours
Measure: Mean (Standard Deviation); unit: second
Arm/Group | Group1 | Group 2 | Group 3 | Group 4 | Group 5 /Control
Number analyzed (Participants) | 34 | 35 | 34 | 36 | 34
second | 279 (189) | 263 (170) | 374 (203) | 247 (183) | 402 (190)

4. Secondary Outcome: Hypoxemia
Description: Check the frequency of hypoxemia episode during induction, procedure, and recovery time
Time Frame: All participants wil be follow for the duration of bronchoscope room stay, an expect average of 2 hours
Measure: Number; unit: participants
Arm/Group | Group1 | Group 2 | Group 3 | Group 4 | Group 5 /Control
Number analyzed (Participants) | 34 | 35 | 34 | 36 | 34
participants
  Induction time | 1 | 9 | 1 | 6 | 1
  Procedure time | 13 | 10 | 16 | 15 | 18
  Recovery time | 5 | 2 | 5 | 4 | 5

5. Secondary Outcome: Hypotension
Description: Check the frequency of hypotension episode during induction, procedure and recovery time
Time Frame: All participants wil be follow for the duration of bronchoscope room stay, an expect average of 2 hours
Measure: Number; unit: participants
Arm/Group | Group1 | Group 2 | Group 3 | Group 4 | Group 5 /Control
Number analyzed (Participants) | 34 | 35 | 34 | 36 | 34
participants
  Induction time | 2 | 1 | 0 | 0 | 0
  Procedure time | 7 | 7 | 11 | 5 | 6
  Recovery time | 4 | 4 | 4 | 2 | 4

ADVERSE EVENTS:
Time Frame: Before, during, and after the fibro-bronchoscopy procedure
Arm/Group | Group1 | Group 2 | Group 3 | Group 4 | Group 5 /Control
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/35 | 0/34 | 0/36 | 0/34
Other Adverse Events (participants affected / at risk) | 0/34 | 0/35 | 0/34 | 0/36 | 0/34

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No